CLINICAL TRIAL: NCT05499364
Title: TinCat Tobacco Cessation Protocol for LGBTQ+ Austinites
Brief Title: TinCat LGBTQ+ Smoking Cessation Via Asynchronous Telehealth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael Parent, Associate professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003092
Record Dates: First submitted 2022-07-24; First posted 2022-08-12 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Tobacco Use Disorder; Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the control or intervention groups randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quit.gov program (Active Comparator): Generic intervention based on quit.gov sessions.
  Interventions: Behavioral: Quit.gov program
- TinCat (Experimental): Individualized asynchronous telehealth including LGBTQ+ affirming components.
  Interventions: Behavioral: TinCat

INTERVENTIONS:
Behavioral: TinCat — 7-10 minute personalized video sessions based in tobacco cessation modules.
  Arms: TinCat
Behavioral: Quit.gov program — 7-10 minute generic videos directing participants through quit.gov program
  Arms: Quit.gov program

SUMMARY:
The purpose of this study is to assess the efficacy of a novel telehealth-based intervention to reduce tobacco use among LGBTQ+ people.

DETAILED DESCRIPTION:
After being informed about potential risks and screened into the study, patients will be randomized into the treatment or control group. Control group participants will complete 7 sessions based on quit.gov smoking cessation planning. Intervention participants will complete 7 sessions of individualized asynchronous telehealth sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Live in Greater Austin
* Identify as LGBTQ+
* Current smokers
* High speed internet access

Exclusion Criteria:

* Exceed screener cutoff for suicide risk
* Exceed screener cutoff for borderline personality disorder
* Report current active substance use other than tobacco that interferes with functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Tobacco use | 11 weeks
  Cigarette and vape assessments based on prior research on vaping/smoking:
  Cigarette: Today, did you have at least one puff on a cigarette (yes/no) IF YES, THEN How many cigarettes did you smoked (at least one puff) (1-"more than 60").
  Vaping: Today, did you use an electronic nicotine delivery system (i.e., a vape containing nicotine), even just one puff? (yes/no) IF YES, THEN How many times they had at least one puff (1 time, 2-5 times, 6-10 times, 11-15 times, 16-20 times, 21-25 times, 26-30 times, 31 or more times).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teah GE, Conner TS. Psychological and Demographic Predictors of Vaping and Vaping Susceptibility in Young Adults. Front Psychol. 2021 Aug 17;12:659206. doi: 10.3389/fpsyg.2021.659206. eCollection 2021. PMID 34484026